CLINICAL TRIAL: NCT05099211
Title: Neuromuscular Deconditioning and Reconditioning in Colon Cancer Patients: A Pilot Study of an APA Muscle Rendorcement Program
Brief Title: Neuromuscular Deconditioning and Reconditioning in Colon Cancer Patients: an APA Muscle Rendorcement Program
Acronym: REMUSCLON
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COTTET CHU Dijon 2018
Record Dates: First submitted 2021-10-12; First posted 2021-10-29 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Colon Cancer; Muscle Strengthening
MeSH Terms: conditions — Colonic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients muscle strengthening (Experimental)
  Interventions: Procedure: Muscle biopsies; Other: Muscle Strengthening; Biological: Blood and urine samples; Other: Evaluation 1 pre-surgery; Other: Evaluation 2 post-surgery; Other: Intermediate Evaluation 3; Other: Final post-training evaluation 4
- Aerobic Training Patients (Experimental)
  Interventions: Procedure: Muscle biopsies; Biological: Blood and urine samples; Other: Aerobic Training; Other: Evaluation 1 pre-surgery; Other: Evaluation 2 post-surgery; Other: Intermediate Evaluation 3; Other: Final post-training evaluation 4
- Healthy patients (Active Comparator)
  Interventions: Biological: Blood and urine samples; Other: Evaluation 1 pre-surgery

INTERVENTIONS:
Procedure: Muscle biopsies — Optional
  In pre-training:
  Biopsy performed during the digestive surgery procedure
  Final evaluation (minimum 1 day and maximum 7 days after the last training session): biopsy performed in the digestive surgery department.
  Arms: Aerobic Training Patients; Patients muscle strengthening
Other: Muscle Strengthening — 3 sessions per week for 18 weeks. Duration: 1 hour Training on different strength training machines for the main muscle groups of the lower and upper limbs. The training load will be gradually increased over the sessions.
  Arms: Patients muscle strengthening
Biological: Blood and urine samples — fasting blood sample taken at assessments 1, 2, 3 and 4 for patients and assessment 1 for controls
Other: Aerobic Training — 3 sessions per week for 18 weeks. Duration: 1 hour Training on a "classic" pedal bicycle (called an ergocycle). The intensity and duration of the training will be gradually increased over the sessions and according to the patient's abilities.
  Arms: Aerobic Training Patients
Other: Evaluation 1 pre-surgery — Carried out at least 15 days before surgery
  1. st visit:
     * Nutritional assessment
     * Body composition
     * Psychometric tests of quality of life + IPAQ Test
     * VO2pic
  2. nd visit:
     * Neuromuscular tests
     * Functional tests
Other: Evaluation 2 post-surgery — 1. st visit:
     * Body composition
     * Nutritional assessment
     * Psychometric tests of quality of life
  2. nd visit:
     * neuromuscular tests
     * Functional tests
     * Familiarization with training equipment if patient participates in re-training
  Arms: Aerobic Training Patients; Patients muscle strengthening
Other: Intermediate Evaluation 3 — performed 9 weeks after the beginning of training Identical tests to evaluation 1 + TM6
  Arms: Aerobic Training Patients; Patients muscle strengthening
Other: Final post-training evaluation 4 — Tests identical to evaluation 1 + TM6
  Arms: Aerobic Training Patients; Patients muscle strengthening

SUMMARY:
Colon cancer is a real public health problem with more than 46,000 new cases diagnosed per year in France and about 650 cases in Burgundy. Muscle deconditioning (MD), which is characterized by a loss of muscle mass and function, is a frequent consequence in cancer patients and conditions the prognosis. Therefore, it is essential to understand its complex etiology in oncology in order to address the real need for therapeutic countermeasures in clinical practice. DM is a multifactorial process that is exacerbated by therapies. It induces neurogenic and muscular alterations that can profoundly affect patients' quality of life.

Currently, analyses of this phenomenon in oncology have been limited essentially to a global evaluation of physical performance, neglecting the muscular and nervous nature of the adaptations responsible for it.

Most studies analyzing the therapeutic effects of physical activity (PA) have shown numerous physiological and psychological benefits of aerobic exercise. However, this form of PA is still not very effective in preserving muscle mass.

Only muscle strengthening can have an anabolic effect by accelerating the rate of protein synthesis.

ELIGIBILITY:
Inclusion Criteria:

* Patient Inclusion Criteria :
* Adult patients who are < 80 years old
* with a first diagnosis of colon cancer, regardless of TNM stage
* to undergo a scheduled excision surgery (laparoscopic colectomy or laparoscopy)
* with WHO stage < 1 to the inclusion visit
* having given their written consent
* living close to the participating center (<50 km)
* ability to understand instructions

Criteria for inclusion of healthy subjects :

* Adult who is < 80 years old
* matched by gender, age and BMI to a patient
* with WHO stage < 1 at visit V1
* no medical contraindications to the program
* having given written consent

Exclusion Criteria:

* Criteria for exclusion of patients and healthy subjects :
* Protected Adult
* Person not affiliated to national health insurance
* Pregnant or breastfeeding woman
* uncontrolled hypertension
* Suffers from unstable diabetes of any type
* Suffers from heart disease. Pre-surgical VO2 test will confirm authorization.
* Affected by any condition likely to complicate the performance of physical activity (neurological, psychiatric, neuromuscular disorders, severe osteoporosis)
* Patient who received neo-adjuvant chemotherapy

Patient-specific exclusion criteria

- Patient with rectal cancer or other evolving cancer

Exclusion criteria specific to healthy subjects

* Subject has had cancer in the last 5 years
* Subject with a high level of physical activity according to the IPAQ questionnaire

Criteria for exclusion of patients and healthy subjects for biopsy:

* Person with keloidosis
* Person with bleeding disorders, and/or on anticoagulant and antiaggregant medication
* hypersensitivity to lidocaine

SECONDARY EXCLUSION CRITERIA FOR TRAINING PATIENTS

* Patient with a WHO stage > 1 at the V2 visit
* Presence of an ostomy (complicates PA practice)
* absence of post-operative chemotherapy treatment
* Refusal of the surgeon and/or oncologist and/or rehabilitation physician to practice PA SECONDARY EXCLUSION CRITERIA FOR HEALTHY SUBJECTS
* subject with a WHO stage > 1 at the V2 visit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the program in terms of the number of sessions attended | Up to Week 30 (evaluation 4) for patients
  Tolerance in terms of level of effort and pain will be tested at each session and will condition the continuation or not of the sessions and therefore acceptability
Acceptability of the program in terms of the number of sessions attended | Up to Week 1 (evaluation 1) for healthy patients
  Tolerance in terms of level of effort and pain will be tested at each session and will condition the continuation or not of the sessions and therefore acceptability

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France